CLINICAL TRIAL: NCT04499014
Title: Evaluation of the Effects of Steroid Phonophoresis and Therapeutic Ultrasound in Carpal Tunnel Syndrome: A Randomized Placebo - Controlled Trial
Brief Title: Ultrasound and Phonophoresis in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir City Hospital (Other)
Responsible Party: Principal Investigator, Fulya Bakılan, Medical Doctor, Eskisehir City Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1234567
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2016-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; steroid phonophoresis; ultrasound
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography; Phonophoresis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ultrasound (Experimental): ultrasound : a frequency of 1 MHz and an intensity of 1 W/cm2, 5 days a week, a total of 10 sessions
  Interventions: Device: ultrasound
- phonophoresis (Experimental): an intensity of 1 W/cm2 and a frequency of 1 MHz and phonophoresis with 0.1% dexamethasone pomade,5 days a week, a total of 10 sessions
  Interventions: Device: ultrasound
- placebo ultrasound (Placebo Comparator): same ultrasound device as described above seemed to be working but without delivering any output, 5 days a week, a total of 10 sessions
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — 5 days a week, a total of 10 sessions
  Other Names: phonophoresis; placebo ultrasound

SUMMARY:
In this placebo-controlled, randomized, prospective study, the efficacy of ultrasonography (US) and steroid phonophoresis (PH) treatments was evaluated in patients with idiopathic carpal tunnel syndrome.

DETAILED DESCRIPTION:
Twenty-seven patients (46 hands) were admitted in this study. Patients were randomly divided three groups. The first group was ultrasound group, the second group was PH group and the third group was placebo US group. Continuous ultrasound with a frequency of 1 MHz, an intensity of 1.0 W/cm2 was used in the US and the PH groups. PH group received 0,1% dexamethasone. Placebo group received a frequency of 0 MHz, an intensity of 0 W/cm² ultrasound. Treatments were administered for 5 days a week, a total of 10 sessions. All patients also wore night splints during treatment. Visual Analogue Scale (VAS), Boston Symptom Severity Scale, Functional Capacity Scale, grip strength and electroneurophysiological evaluations were compared before the treatment, after the treatment and three months later.

ELIGIBILITY:
Inclusion Criteria:

* Mild or moderate idiopathic carpal tunnel syndrome (without thenar atrophy or spontaneous activity on electrophysiological examination of the abductor pollicis brevis (APB) muscle)

Exclusion Criteria:

* The patients with medical problems (diabetes mellitus, hypothyroidism, rheumatic diseases, acute trauma, pregnancy etc.)
* cervical radiculopathy
* etiologic factors which predispose to or polyneuropathy
* reinnervation or fibrillation potentials in their abductor pollicis brevis muscles
* physical or medical therapy within 3 months for CTS and steroid injection applied
* experience CTS median nerve trauma and CTS surgery
* serious thenar atrophy and anesthesia
* contraindication in steroid treatment (steroid allergies, hypertension etc.)
* contraindication in ultrasonic therapy (bleeding disorders, acute inflammation of the joints, acute infections, cancer and precancerous lesions, arteriovenous circulatory disorders etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2016-01-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | three month
  Change from baseline in pain with Visual Analogue Scale:Patients were asked to express the pain felt by them using 0-10 scales, 0 no pain and 10 the most severe pain faced throughout their life.
Boston Symptom Severity Scale | three month
  Change from baseline in symptom severity with Boston Symptom Severity Scale:Patients were asked to choose an answer among five answers taking 1- 5 points in the questionnaires with 11 statements. Total point was divided into the number of statements and the score was determined and high scores were interpreted as increased symptom severity
Boston Functional Capacity Scale | three month
  Change from baseline in functional status with Boston Functional Capacity Scale:Patients were asked to choose an answer among five answers taking 1- 5 points in the questionnaires with 11 statements. Total point was divided into the number of statements and average score was determined and high scores were interpreted as functionality deformation in the hands
grip strength | three month
  Change from baseline in strength with grip strength:To assess the grip strength, baseline hydraulic hand dynamometer was used. 3 measurements were made for each patient and the average of them was calculated
electroneurophysiological evaluations | three month
  Change from baseline electroneurophysiological measurement:The median nerve motor conduction velocity(m/s) , the median nerve motor distal latency(ms), 2nd finger - palm median nerve sensory distal latency(ms), 2nd finger - palm median nerve sensory conduction velocity(m/s), median sensory nerve conduction velocity(m/s) and median nerve sensory distal latency between the wrist and palm(ms)

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Ortanca, Principal Investigator — Eskişehir City Hospital